CLINICAL TRIAL: NCT05831865
Title: The Efficacy and Safety of Autologous Stem Cell Transplantation (ASCT) in Frontline Therapy of Patients With High-Risk Diffuse Large B-Cell Lymphoma
Brief Title: Frontline of ASCT in High-risk DLBCL
Acronym: Essential
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, JinLu, Professor of Medicine and Hematology, Deputy Director of the Department of Hematology, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2023PHB119
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: autologous stem cell transplantation; international prognostic index
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DLBCL patients achieving CR or CMR during interim evaluation: During the interim evaluation, patients achieving complete response (CR) as determined by computed tomography (CT), or complete metabolic response (CMR) as determined by positron emission tomography-computed tomography (PET-CT), will be followed up for up to two years after completing the R-CHOP regimen followed by ASCT.
- DLBCL patients achieving PR or PMR during interim evaluation: During the interim evaluation, patients achieving partial response (PR) as determined by CT, or partial metabolic response (PMR) as determined by PET-CT, and who are willing to receive Pola-R-CHP as the following treatment regimen followed by ASCT with Pola-BEAM as conditioning regimen, will also be followed up for up to two years.

SUMMARY:
The role of frontline therapy of autologous stem cell transplant (ASCT) in diffuse large B-cell lymphoma (DLBCL) is controversial. The investigators aim to conduct this prospective study to observe the efficacy and safety of ASCT as frontline therapy in DLBCL patients with high-risk disease, defined by an International Prognostic Index (IPI) score equal to or greater than three.

DETAILED DESCRIPTION:
There is evidence to suggest that chemotherapy followed by ASCT may be more effective than standard chemotherapy alone as a frontline treatment for high-risk DLBCL patients. However, the use of ASCT as frontline therapy for DLBCL remains controversial due to concerns over the potential toxicities of the procedure, as well as questions about which patients would benefit most from this approach.

The investigators aim to conduct this prospective study to observe the efficacy and safety of ASCT as frontline therapy in DLBCL patients with high-risk disease, defined by an International Prognostic Index (IPI) score equal to or greater than 3 points.

Patients diagnosed with DLBCL and an IPI score of equal to or greater than three will be eligible for inclusion in this study, provided they consent to receive the standard R-CHOP (Rituximab, cyclophosphamide, hydroxydaunomycin, oncovin, and prednisone) regimen, followed by ASCT. During the interim evaluation, patients achieving complete response (CR) as determined by computed tomography (CT), or complete metabolic response (CMR) as determined by positron emission tomography-computed tomography (PET-CT), will be followed up for up to two years after completing the R-CHOP regimen followed by ASCT. Patients achieving partial response (PR) as determined by CT, or partial metabolic response (PMR) as determined by PET-CT, and who are willing to receive Pola-R-CHP (Polatuzumab vedotin, rituximab, cyclophosphamide, hydroxydaunomycin, and prednisone) as the following treatment regimen followed by ASCT with Pola-BEAM (Polatuzumab vedotin, carmustine/bendamustine, etoposide, cytarabine and melphalan) as conditioning regimen, will also be followed up for up to two years. Patients achieving less than a PR or PMR response will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated participants with cluster of differentiation 20 (CD20)-positive DLBCL, including one of the following diagnoses by 2016 World Health Organization (WHO) classification of lymphoid neoplasms: DLBCL, not otherwise specified (NOS) including germinal center B-cell type, activated B-cell type; T-cell/histiocyte-rich large B-cell lymphoma; Epstein-Barr virus-positive DLBCL, NOS; anaplastic lymphoma kinase (ALK)-positive large B-cell lymphoma; human herpesvirus-8 (HHV8)-positive DLBCL, NOS; High-grade B-cell lymphoma with MYC and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements (double-hit or triple-hit lymphoma); High-grade B-cell lymphoma, NOS
* Measurable tumor assessed by Lugano Response Criteria
* International Prognostic Index (IPI) score equal to or greater than 3 points
* Adequate hematologic function
* Adequate liver function
* Adequate kidney function
* Left ventricular ejection fraction (LVEF) >/= 50 percent (%) on cardiac echocardiogram (ECHO)

Exclusion Criteria:

* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* Participants with central nervous system (CNS) lymphoma (primary or secondary involvement)
* History of other malignancy that could affect compliance with the protocol or interpretation of results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with DLBCL and an IPI score equal to or greater than three and consent to receive the standard R-CHOP regimen followed by ASCT. During the interim evaluation, patients achieving CR or CMR, will be followed up for up to two years after completing the R-CHOP regimen followed by ASCT. Patients achieving PR or PMR and who are willing to receive Pola-R-CHP as the following treatment regimen followed by ASCT, will also be followed up for up to two years. Patients achieving less than a PR or PMR response will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-04-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  From the start of treatment to the first occurrence of disease progression or relapse, or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Percentage of Participants With complete response (CR) or complete metabolic response (CMR) | 2 years
  Assessed by Lugano Response Criteria
Percentage of Participants With partial response (PR) or partial metabolic response (PMR) | 2 years
  Assessed by Lugano Response Criteria
Overall survival (OS) | 2 years
  From the start of treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No